CLINICAL TRIAL: NCT04174027
Title: The Effect of Perturbration on Balance Control in Adults
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MeirMc102-19CTIL
Record Dates: First submitted 2019-10-03; First posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Chronic Ankle Instability
Keywords: Chronic ankle instability ( CAI ); Perturbration; reactive postural control; balance; center of pressure - COP

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Balance control in respond to an unexpected platform perturbration during standing and walking: comparison between individuals with chronic ankle instability and healthy individuals.

DETAILED DESCRIPTION:
An unexpected postural perturbration is a major risk factor of falls and injuries during gait. A postural perturbration is a sudden change in conditions that displaces the body posture away from equilibrium. Reactive postural control response is an immediate ( 70-120 ms ) automatic "like reflex" response which is initiated by unexpected postural perturbration in order to maintain balance. Even among young healthy adults there could be a problem in balance performance which does not become evident untill a slip or a trip or any other sudden perturbration happens. Thus a simple test of pertubration while standing or walking can identify a problem .

This study is comparing the reactive postural control of physical education students who suffer from chronic ankle instability (CAI) to healthy students on a Perturbation Treadmill. The device consists of a treadmill mounted on a moving force plate platform. The platform moves in the medial/ lateral plains to simulate a slip and a trip in both the standing and walking phase. Their reactive postural control is tested in a few conditions: standing on both legs - eyes open and eyes closed, in tandem standing, standing on one leg and in walking. In each condition the perturbration is given every 5-15 seconds in different speed and in unexpected direction (right /left). Lost of balance control is any change in the original location of the foot in standing conditions or stepping out of the treadmill.

ELIGIBILITY:
Inclusion Criteria:

* age 18-50
* good health
* active people

Exclusion Criteria:

* Body weight greater than 135 kg
* Bone instability (non-consolidated fractures, unstable spinal column, severe osteoporosis)
* Head damage in the year prior to the study
* Diabetics or Unstable circulation
* Cardiac (blood) contraindications
* Vestibular problem
* Neurological deficits
* Mechanical ventilation problem
* Severe vascular disorders of the lower limbs

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Physical education students from Zinman College in Wingate
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-12-15 (Estimated); Primary Completion 2020-10-15 (Estimated); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
static balance control in reaction to perturbration | 20 minutes
  The angle velocity at the ankle at the moment of loosing postural control while standing
dynamic balance control un reaction to perturbration | 10 minutes
  the speed of perturbration at the moment of loosing balance while walking

SECONDARY OUTCOMES:
Time to returning to original condition | 30 minutes
  How much time it takes to come back to the original step (Center of Pressure - COP) after the perturbration

OTHER OUTCOMES:
movement inside the foot during balance control. | 30 minutes
  The changes in center of pressure (COP) amplitude height

IPD SHARING:
Plan to Share IPD: No